CLINICAL TRIAL: NCT03364738
Title: An Open-label Study Investigating the Safety and Efficacy of rhPTH(1-84) in Subjects With Hypoparathyroidism
Brief Title: Safety and Efficacy Study of rhPTH(1-84) in Subjects With Hypoparathyroidism
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to Takeda commercial Natpara recall.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP634-404; 2017-003067-36 (EudraCT Number)
Record Dates: First submitted 2017-11-20; First posted 2017-12-07 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2021-05

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rhPTH(1-84) (Experimental): Participants will receive rhPTH(1-84) subcutaneous (SC) injection in the thigh (alternate thigh every day) once daily (QD) of an escalating dose from 50 microgram (mcg) to a maximum of 100 mcg increased in increments of 25 mcg no more frequently than every 2 to 4 weeks, with the goal of achieving or maintaining albumin-corrected serum calcium (ACSC) levels in the range of 2-2.25 millimoles per liter (mmol/L) (8.0-9.0 milligrams per deciliter [mg/dL]). Once a participant achieves a stable ACSC (2-2.25 mmol/L [8.0-9.0mg/dL]) and has minimized supplement doses, they will be maintained at that dose of rhPTH(1-84). If ACSC is greater than (>) 2.25 mmol/L (>9.0 mg/dL), a starting dose of 25 mcg will be administered.
  Interventions: Biological: rhPTH(1-84)

INTERVENTIONS:
Biological: rhPTH(1-84) — Participants will receive rhPTH(1-84) SC injection in the thigh (alternate thigh every day) QD.

SUMMARY:
This study is open to adults with hypoparathyroidism who complete the SHP634-101 study (PARALLAX Study). The purpose of this study is to see if rhPTH(1-84) is safe and effective in adults with hypoparathyroidism who previously participated in the SHP634-101 study. All participants enrolled in this study will receive rhPTH(1-84) once-daily for 52 weeks via an injection.

Patients who complete the SHP634-101 study will have the option to screen for this extension study.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions
* Ability to voluntarily provide written, signed, and dated informed consent to participate in the study.
* Previously completed the SHP634-101 (NCT02781844) study, including the 30-day follow-up.
* Male or non-pregnant, non-lactating female subjects who agree to comply with applicable contraceptive requirements of the protocol or females of non-childbearing potential.

Exclusion Criteria:

* Received investigational study drug, aside from that received in study SHP634-101 (NCT02781844), within 3 months prior to the screening visit.
* Presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine (with exception of the condition under study), or neurologic system(s) or psychiatric disease, that in the opinion of the investigator, would make the subject unsuitable for this study.
* Received parathyroid hormone (PTH), PTH analog, or parathyroid hormone fragment 1-34 [PTH(1-34)] treatment within the last 30 days from the screening visit.
* Subjects with a history of parathyroid hormone intolerance, based on investigator determination.
* Any disease that might affect calcium metabolism or calcium-phosphate homeostasis as determined by the investigator other than hypoparathyroidism, including but not limited to, active hyperthyroidism; poorly controlled insulin-dependent diabetes mellitus or type 2 diabetes mellitus; severe and chronic cardiac, liver or renal disease; Cushing's syndrome; neuromuscular disease such as rheumatoid arthritis; myeloma; pancreatitis; malnutrition; rickets; recent prolonged immobility; active malignancy, bone metastases or a history of skeletal malignancies; primary or secondary hyperparathyroidism; a history of parathyroid carcinoma; hypopituitarism, acromegaly; or multiple endocrine neoplasia types 1 and 2 .
* Subjects who are at increased baseline risk for osteosarcoma such as subjects with Paget's disease of bone or unexplained elevations of alkaline phosphatase, young adult subjects with open epiphyses, subjects with hereditary disorders predisposing to osteosarcoma or subjects with a prior history of external beam or implant radiation therapy involving the skeleton.
* Use of the following medications prior to administration of investigational product within:

  1. 30 days-loop diuretics, lithium, systemic corticosteroids (medical judgment is required by the investigator. Primarily high doses of systemic corticosteroids [example (eg), prednisone] should be excluded. Stable doses of hydrocortisone [eg, as treatment for Addison's disease] may be acceptable).
  2. 3 months-cinacalcet hydrochloride
  3. 6 months-fluoride tablets, oral bisphosphonates, methotrexate, growth hormone, digoxin
  4. 12 months-intravenous bisphosphonates, drug or alcohol abuse, as determined by the investigator
* Presence of any clinically significant results from laboratory tests, vital signs assessments, or electrocardiograms (ECG), that in the opinion of the investigator, would make the subject unsuitable for this study.
* Any medical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for this study.
* History of a clinically significant illness during the 4 weeks prior to dosing, that in the opinion of the investigator, would make the subject unsuitable for this study.
* History of any clinically significant surgery or procedure within 8 weeks of first dose, as determined by the investigator or expected to undergo a major surgical procedure during the trial.
* History of an allergic response(s) to PTH, PTH analogs, or PTH(1-34), or other clinically significant allergies, that in the opinion of the investigator, would make the subject unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (10):
- United States (5):
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Crescent City Clinical Research Center, LLC, Metairie, Louisiana
  - Northern Nevada Endocrinology - Lisa Abbott MD, Reno, Nevada
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Jefferson Rheumatology Associates, Philadelphia, Pennsylvania
- Canada (2):
  - Bone Research and Education Centre, Oakville, Ontario
  - CHU de Quebec-Universite Laval, Québec
- Aarhus Universitetshospital, Aarhus N, Denmark
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Pecsi Tudomanyegyetem, I. sz. Belgyogyaszati Klinika, Pécs

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Khan AA, Abbott LG, Ahmed I, Ayodele O, Gagnon C, Finkelman RD, Mezosi E, Rejnmark L, Takacs I, Yin S, Ing SW. Open-label extension of a randomized trial investigating safety and efficacy of rhPTH(1-84) in hypoparathyroidism. JBMR Plus. 2024 Jan 5;8(3):ziad010. doi: 10.1093/jbmrpl/ziad010. eCollection 2024 Mar. PMID 38741607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hypoparathyroidism (HPT) who completed SHP634-101 (NCT02781844) study were eligible and enrolled in this extension study which was conducted at 10 sites in the United States, Denmark, Hungary and Canada between 26 September 2018 (first participant first visit) and 14 April 2020 (last participant last visit).
Pre-assignment Details: A total of 22 participants were enrolled and treated in the study, of which 14 participants completed the study.
Groups:
- rhPTH(1-84): Participants received recombinant human parathyroid hormone (rhPTH) (1-84) (Natpara) 50 microgram (mcg), injection, subcutaneously, once daily in the thigh (alternate thigh every day) up to 52 weeks (end of treatment [EOT])/ early termination (ET). Dose escalation was done up to 100 mcg in increments of 25 mcg no more frequently than every 2 to 4 weeks, with the goal of achieving or maintaining albumin-corrected serum calcium (ACSC) levels in the range of 2-2.25 millimoles per liter (mmol/L) (8-9 milligrams per deciliter [mg/dL]). Administered dose was maintained once a participant achieved a stable ACSC level of 2-2.25 mmol/L (8-9 mg/dL) and had minimized supplement (active vitamin D and calcium supplement) doses. If ACSC was greater than (>) 2.25 mmol/L (>9.0 mg/dL), a starting dose of 25 mcg was administered.
Period: Overall Study
Arm/Group | rhPTH(1-84)
Started | 22
Completed | 14
Not Completed | 8
Not completed — Early termination due to Food and Drug Administration recall of rhPTH(1-84) (Natpara) | 6
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis population consisted of all participants who have received at least 1 dose of rhPTH(1-84).
Groups:
- rhPTH(1-84): Participants received rhPTH(1-84) (Natpara) 50 mcg, injection, subcutaneously, once daily in the thigh (alternate thigh every day) up to 52 weeks (EOT/ET). Dose escalation was done up to 100 mcg in increments of 25 mcg no more frequently than every 2 to 4 weeks, with the goal of achieving or maintaining ACSC levels in the range of 2-2.25 mmol/L (8-9 mg/dL). Administered dose was maintained once a participant achieved a stable ACSC level of 2-2.25 mmol/L (8-9 mg/dL) and had minimized supplement (active vitamin D and calcium supplement) doses. If ACSC was >2.25 mmol/L (>9.0 mg/dL), a starting dose of 25 mcg was administered.
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 1
  White | 20
  Native Hawaiian or other Pacific Islander | 0
  Native American And Caucasian | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Total Albumin-corrected Serum Calcium (ACSC) Values Greater Than or Equal to (>=) to the Range of 7.5 mg/dL (1.875 mmol/L) and Less Than or Equal to (<=) Upper Limit of Normal (ULN) at Week 24
Description: Percentage of participants who achieved ACSC values >= to range of 1.875 mmol/L and <= ULN at Week 24 was reported.
Time Frame: At Week 24
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84). Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 21
percentage of participants | 100

2. Primary Outcome: Percentage of Participants With Total ACSC Values >= to the Range of 7.5 mg/dL (1.875 mmol/L) and <=ULN at Week 52 (End-of-treatment [EOT])
Description: Percentage of participants who achieved ACSC values >= to range of 1.875 mmol/L and <= ULN at Week 52 (EOT) was reported.
Time Frame: At Week 52 (EOT)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84).
Measure: Number; unit: percentage of participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
percentage of participants | 95.5 [0.772 to 0.999]

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A Serious Adverse Event (SAE) was any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect, and is an important medical event. TEAEs were defined as AEs with a start date on or after the first dose of investigational product or a start date before the date of the first dose of investigational product that increased in severity or after the date of the first dose.
Time Frame: From start of study drug administration to end of study (Week 56)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
Participants
  Participants with TEAEs | 17
  Participants with serious TEAEs | 4

4. Primary Outcome: Number of Participants With Clinically Significant Change in Clinical Laboratory Values
Description: Clinical laboratory assessment included hematology, serum chemistry, urine chemistry and urinalysis. Clinical significance was judged by the investigator based upon the out of range values of standard range set for each parameter. Any changes in clinical laboratory results which were deemed clinically significant by the investigator was reported.
Time Frame: From start of study drug administration to end of study (Week 56)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
Participants | 0

5. Primary Outcome: Number of Participants With Clinically Significant Change in Vital Sign
Description: Vital sign parameters included: temperature, pulse rate, respiration rate, systolic and diastolic blood pressure. Clinical significance was judged by the investigator based upon the out of range values of standard range set for each parameter. Any changes in vital signs which were deemed clinically significant by the investigator was reported.
Time Frame: From start of study drug administration to end of study (Week 56)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Groups:
- rhPTH(1-84): Participants received rhPTH(1-84) (Natpara) 50 mcg, injection, subcutaneously, once daily in the thigh (alternate thigh every day) up to 52 weeks (EOT])/ET). Dose escalation was done up to 100 mcg in increments of 25 mcg no more frequently than every 2 to 4 weeks, with the goal of achieving or maintaining ACSC levels in the range of 2-2.25 mmol/L (8-9 mg/dL). Administered dose was maintained once a participant achieved a stable ACSC level of 2-2.25 mmol/L (8-9 mg/dL) and had minimized supplement (active vitamin D and calcium supplement) doses. If ACSC was >2.25 mmol/L (>9.0 mg/dL), a starting dose of 25 mcg was administered.
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
Participants | 0

6. Primary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Parameters
Description: Twelve-lead ECGs was performed in triplicate with a minimum 2-minute gap between traces. The participant rested in the supine position for at least 5 minutes before collecting the ECG. Assessment of ECG parameters included: heart rate, RR interval, PR interval, QRS interval, QT interval, and QTc interval. Clinical significance was judged by the investigator based upon the out of range values of standard range set for each parameter. Any change in ECG assessments which were deemed clinically significant by the investigator was reported.
Time Frame: From start of study drug administration to end of study (Week 56)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
Participants | 0

7. Primary Outcome: Number of Participants With Clinically Significant Change in Estimated Glomerular Filtration Rate (eGFR) Values
Description: eGFR was calculated using the chronic kidney disease epidemiology (CDK-epi) formula. Clinical significance was judged by the investigator based upon the out of range values of standard range set for parameter. Any change in eGFR assessments which were deemed clinically significant by the investigator was reported.
Time Frame: From start of study drug administration to end of study (Week 56)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
Participants | 0

8. Primary Outcome: Number of Participants With Clinically Significant Change in Serum Creatinine Value
Description: eGFR was assessed by measuring serum creatinine. Serum creatinine level was obtained directly from laboratory results. Clinical significance was judged by the investigator based upon the out of range values of standard range set for parameter. Any change in serum creatinine assessments which were deemed clinically significant by the investigator was reported.
Time Frame: From start of study drug administration to end of study (Week 56)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
Participants | 0

9. Primary Outcome: Number of Participants With Positive Anti-Parathyroid Hormone Antibodies at Week 24
Description: Number of participants with positive anti-parathyroid hormone antibodies at Week 24 was reported.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 21
Participants | 0

10. Secondary Outcome: Change From Baseline in Albumin Corrected Serum Calcium (ACSC) Concentration at Weeks 24 and 52 (EOT)
Description: Change from baseline in ACSC concentration at Weeks 24 and 52 (EOT) was reported.
Time Frame: Baseline, Weeks 24 and 52 (EOT)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84). Here "number analyzed" were participants who were evaluable for the outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
mmol/L
  Change at Week 24: number analyzed (Participants) | 21
  Change at Week 24 | -0.024 (0.2065)
  Change at Week 52 (EOT) | -0.076 (0.1497)

11. Secondary Outcome: Change From Baseline in Serum Phosphate Concentration at Weeks 4, 8, 16, 24, 32, 40 and 52 (EOT)
Description: Change from baseline in serum phosphate concentration at Weeks 4, 8, 16, 24, 32, 40 and 52 (EOT) was reported.
Time Frame: Baseline, Weeks 4, 8, 16, 24, 32, 40 and 52 (EOT)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
mmol/L
  Change at Week 4: number analyzed (Participants) | 21
  Change at Week 4 | -0.167 (0.1816)
  Change at Week 8: number analyzed (Participants) | 21
  Change at Week 8 | -0.124 (0.2252)
  Change at Week 16: number analyzed (Participants) | 21
  Change at Week 16 | -0.107 (0.2583)
  Change at Week 24: number analyzed (Participants) | 21
  Change at Week 24 | -0.160 (0.2303)
  Change at Week 32: number analyzed (Participants) | 20
  Change at Week 32 | -0.089 (0.1809)
  Change at Week 40: number analyzed (Participants) | 17
  Change at Week 40 | -0.121 (0.2542)
  Change at Week 52 (EOT) | -0.114 (0.2590)

12. Secondary Outcome: Change From Baseline in ACSC-phosphate Product at Weeks 4, 8, 16, 24, 32, 40 and 52 (EOT)
Description: Change from baseline in ACSC-phosphate product at Weeks 4, 8, 16, 24, 32, 40 and 52 (EOT) was reported. Here "mmol^2/L^2" is abbreviated as millimoles square per liter square.
Time Frame: Baseline, Weeks 4, 8, 16, 24, 32, 40 and 52 (EOT)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmol^2/L^2
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
mmol^2/L^2
  Change at Week 4: number analyzed (Participants) | 21
  Change at Week 4 | -0.31 (0.462)
  Change at Week 8: number analyzed (Participants) | 21
  Change at Week 8 | -0.19 (0.537)
  Change at Week 16: number analyzed (Participants) | 21
  Change at Week 16 | -0.16 (0.609)
  Change at Week 24: number analyzed (Participants) | 21
  Change at Week 24 | -0.38 (0.556)
  Change at Week 32: number analyzed (Participants) | 20
  Change at Week 32 | -0.29 (0.456)
  Change at Week 40: number analyzed (Participants) | 17
  Change at Week 40 | -0.29 (0.572)
  Change at Week 52 (EOT) | -0.34 (0.539)

13. Secondary Outcome: Change From Baseline in 24-hour Urine Calcium Excretion at Weeks 16, 32 and 52 (EOT)
Description: Change from baseline in 24-hour urine calcium excretion at Weeks 16, 32 and 52 (EOT) was reported.
Time Frame: Baseline, Weeks 16, 32 and 52 (EOT)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84). Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure and "number analyzed" were participants who were evaluable for the outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: millimoles per day (mmol/day)
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 21
millimoles per day (mmol/day)
  Change at Week 16 | -0.22 (4.741)
  Change at Week 32: number analyzed (Participants) | 20
  Change at Week 32 | -3.13 (4.103)
  Change at Week 52 (EOT): number analyzed (Participants) | 20
  Change at Week 52 (EOT) | -2.53 (4.421)

14. Secondary Outcome: Percentage Change From Baseline in Prescribed Supplemental Oral Calcium Dose at Weeks 4, 8, 16, 24, 32, 40, 52 (EOT) and 56 (End of Study [EOS])
Description: Percentage change from baseline in prescribed supplemental oral calcium dose at Weeks 4, 8, 16, 24, 32, 40, 52 (EOT) and 56 (EOS) were reported.
Time Frame: Baseline and at Weeks 4, 8, 16, 24, 32, 40, 52 (EOT) and 56 (EOS)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84). Here "number analyzed" were participants who were evaluable for the outcome measure at given time points. Data for Week 56 was not collected as study was early terminated due to FDA recall of rhPTH(1-84) (Natpara).
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
percentage change
  Percentage change at Week 4: number analyzed (Participants) | 21
  Percentage change at Week 4 | -14.30 (34.269)
  Percentage change at Week 8: number analyzed (Participants) | 21
  Percentage change at Week 8 | -29.08 (38.019)
  Percentage change at Week 16: number analyzed (Participants) | 21
  Percentage change at Week 16 | -36.94 (45.665)
  Percentage change at Week 24: number analyzed (Participants) | 21
  Percentage change at Week 24 | -49.05 (49.049)
  Percentage change at Week 32: number analyzed (Participants) | 20
  Percentage change at Week 32 | -55.58 (44.268)
  Percentage change at Week 40: number analyzed (Participants) | 17
  Percentage change at Week 40 | -56.36 (45.168)
  Percentage change at Week 52 (EOT) | -48.55 (45.237)
  Percentage change at Week 56 (EOS): number analyzed (Participants) | 0

15. Secondary Outcome: Percentage Change From Baseline in Prescribed Supplemental Active Vitamin D Dose at Weeks 4, 8, 16, 24, 32, 40, 52 (EOT) and 56 (EOS)
Description: as for outcome 14
Time Frame: Baseline, Weeks 4, 8, 16, 24, 32, 40, 52 (EOT) and 56 (EOS)
Population: Safety analysis population consisted of all participants who had received at least 1 dose of rhPTH(1-84). Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure and "number analyzed" were participants who were evaluable for the outcome measure at given time points. Data for Week 56 was not collected as study was early terminated due to FDA recall of rhPTH(1-84) (Natpara).
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 21
percentage change
  Percentage change at Week 4: number analyzed (Participants) | 20
  Percentage change at Week 4 | -57.50 (40.995)
  Percentage change at Week 8: number analyzed (Participants) | 20
  Percentage change at Week 8 | -70.00 (39.217)
  Percentage change at Week 16: number analyzed (Participants) | 20
  Percentage change at Week 16 | -80.83 (27.185)
  Percentage change at Week 24: number analyzed (Participants) | 20
  Percentage change at Week 24 | -85.42 (25.055)
  Percentage change at Week 32: number analyzed (Participants) | 19
  Percentage change at Week 32 | -90.79 (17.324)
  Percentage change at Week 40: number analyzed (Participants) | 16
  Percentage change at Week 40 | -90.10 (18.564)
  Percentage change at Week 52 (EOT) | -77.38 (43.870)
  Percentage change at Week 56 (EOS): number analyzed (Participants) | 0

16. Secondary Outcome: Percentage Change From Baseline in Serum Bone-specific Alkaline Phosphatase at Weeks 8, 24 and 52 (EOT)
Description: Percentage change from baseline in serum bone-specific alkaline phosphatase at Weeks 8, 24 and 52 (EOT) was reported.
Time Frame: Baseline, Weeks 8, 24 and 52 (EOT)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
percentage change
  Percentage change at Week 8: number analyzed (Participants) | 20
  Percentage change at Week 8 | 29.90 (31.575)
  Percentage change at Week 24: number analyzed (Participants) | 21
  Percentage change at Week 24 | 89.14 (54.452)
  Percentage change at Week 52 (EOT) | 94.08 (75.066)

17. Secondary Outcome: Percentage Change From Baseline in Serum Osteocalcin at Weeks 8, 24 and 52 (EOT)
Description: Percentage change from baseline in serum osteocalcin at Weeks 8, 24 and 52 (EOT) was reported.
Time Frame: Baseline, Weeks 8, 24 and 52 (EOT)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
percentage change
  Percentage change at Week 8: number analyzed (Participants) | 21
  Percentage change at Week 8 | 61.74 (68.363)
  Percentage change at Week 24: number analyzed (Participants) | 21
  Percentage change at Week 24 | 225.91 (130.798)
  Percentage change at Week 52 (EOT) | 294.93 (215.100)

18. Secondary Outcome: Percentage Change From Baseline in Procollagen 1 N-Terminal Propeptide at Weeks 8, 24 and 52 (EOT)
Description: Percentage change from baseline in procollagen 1 N-terminal propeptide at Weeks 8, 24 and 52 (EOT) was reported.
Time Frame: Baseline, Weeks 8, 24 and 52 (EOT)
Population: as for outcome 10
Measure: Median (Standard Deviation); unit: percentage change
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
percentage change
  Percentage change at Week 8: number analyzed (Participants) | 21
  Percentage change at Week 8 | 119.98 (161.156)
  Percentage change at Week 24: number analyzed (Participants) | 21
  Percentage change at Week 24 | 412.46 (248.423)
  Percentage change at Week 52 (EOT) | 476.07 (377.383)

19. Secondary Outcome: Percentage Change From Baseline in Type I Collagen C-Telopeptides at Weeks 8, 24 and 52 (EOT)
Description: Percentage change from baseline in type I collagen C-telopeptides at Week 8, 24 and 52 (EOT) was reported.
Time Frame: Baseline, Weeks 8, 24 and 52 (EOT)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
percentage change
  Percentage change at Week 8: number analyzed (Participants) | 21
  Percentage change at Week 8 | 124.62 (160.564)
  Percentage change at Week 24: number analyzed (Participants) | 21
  Percentage change at Week 24 | 254.26 (198.947)
  Percentage change at Week 52 (EOT) | 227.13 (182.262)

20. Secondary Outcome: Percentage Change From Baseline in Type I Collagen N-Telopeptides at Weeks 8, 24 and 52 (EOT)
Description: Percentage change from baseline in type I collagen N-telopeptides at Week 8, 24 and 52 (EOT) was reported.
Time Frame: Baseline, Weeks 8, 24 and 52 (EOT)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 22
percentage change
  Percentage change at Week 8: number analyzed (Participants) | 21
  Percentage change at Week 8 | 71.33 (99.933)
  Percentage change at Week 24: number analyzed (Participants) | 21
  Percentage change at Week 24 | 183.23 (160.350)
  Percentage change at Week 52 (EOT) | 231.80 (270.229)

21. Primary Outcome: Number of Participants With Positive Anti-Parathyroid Hormone Antibodies at Week 52 (EOT)
Description: Number of participants with positive anti-parathyroid hormone antibodies at Week 52 (EOT) was reported.
Time Frame: Week 52 (EOT)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH(1-84)
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: From start of screening up to end of study (Week 56)
Arm/Group | rhPTH(1-84)
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 10/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhPTH(1-84) (N=22)
Appendicitis (Infections and infestations) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhPTH(1-84) (N=22)
Nausea (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 2 (4)
Fatigue (General disorders) | 4 (5)
Nasopharyngitis (Infections and infestations) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (7)
Migraine (Nervous system disorders) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated due to Takeda commercial Natpara recall.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT03364738/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT03364738/SAP_001.pdf